CLINICAL TRIAL: NCT00441350
Title: Phase III Study Evaluating the Efficacy and Safety of Olmesartan Medoxomil/Hydrochlorothiazide 40/12.5 mg Combination Therapy Versus Olmesartan Medoxomil 40 mg Monotherapy in Patients With Essential Hypertension
Brief Title: Olmesartan/HCTZ 40/12.5 mg Combination Therapy Versus Olmesartan Medoxomil 40 mg Monotherapy in Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menarini Group (Industry)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS866CM-B-E303
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2009-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OM 40 (Active Comparator): Olmesartanmedoxomil (OM)40 mg tablets.
  Interventions: Drug: OM 40
- OM/HCTZ 40/12.5 (Experimental): Olmesartanmedoxomil (OM) /Hydrochlorothiazide (HCTZ)40/12.5 mg tablets.
  Interventions: Drug: OM/HCTZ 40/12.5

INTERVENTIONS:
Drug: OM 40 — Initially patients were to be treated with Olmesartanmedoxomil (OM)40 mg tablets once daily for 8 weeks. After 8 weeks non-responders were to be uptitrated to OM/HCTZ 40/12.5 mg and responders remained on the previous therapy for further 8 weeks.
  Other Names: Treatment
  Arms: OM 40
Drug: OM/HCTZ 40/12.5 — Initially patients were to be treated with Olmesartanmedoxomil (OM) /Hydrochlorothiazide (HCTZ)40/12.5 mg tablets once daily for 8 weeks. After 8 weeks non-responders were to be uptitrated to OM/HCTZ 40/25 mg and responders remained on the previous therapy for further 8 weeks.
  Other Names: Treatment
  Arms: OM/HCTZ 40/12.5

SUMMARY:
The primary objective of this study was to assess the anti-hypertensive effect of OM/HCTZ 40/12.5 mg combination therapy compared to OM 40 mg monotherapy in lowering sitting diastolic BP in hypertensive patients after 8 weeks of double-blind treatment.

The study consisted of two sequential phases of 8 weeks duration each:

During the first phase, OM 40 mg monotherapy was compared with OM/HCTZ 40/12.5 mg in order to evaluate the additional benefit of OM/HCTZ 40/12.5 mg in the treatment of essential moderate to severe hypertension.

During the second phase, patients whose BP proved to be insufficiently controlled by the OM 40 mg monotherapy were to start OM/HCTZ 40/12.5 mg combination therapy while patients whose BP proved to be insufficiently controlled by the OM/HCTZ 40/12.5 mg combination were to be up-titrated to the OM/HCTZ 40/25 mg combination to evaluate the additional benefit of the up-titrated combination.

The study was be conducted by qualified and experienced personnel with adherence to GCP, current guidelines on the design of studies in hypertension, the applicable regulatory requirements and the ethical principles based on the Declaration of Helsinki.

DETAILED DESCRIPTION:
Methodology:

After the signature of the informed consent, patients were screened for eligibility and eligible patients entered into a pre-randomisation period consisting of a taper-off phase of approximately 1-2 weeks (during which patients treated for hypertension were to discontinue their antihypertensive therapy) followed by a 2-week single-blind placebo run-in phase (Visit 1). After conclusion of the placebo run-in phase (Visit 2), eligible patients were randomised to the double-blind active treatment period which consisted of two phases:

First double-blind treatment phase (Phase A, from Randomisation to Week 8):

Eligible patients with mean sitting sBP ≥ 160 and ≤ 200 mmHg and dBP ≥ 100 mmHg and ≤ 120 mmHg were randomised in a 1:2 ratio to receive either OM 40 mg or OM/HCTZ 40/12.5 mg for a total of 8 weeks of treatment (Phase A). Study visits were held after 4 and 8 weeks of double-blind active treatment (Visit 3 and 4, respectively). After 8 weeks (Visit 4), patients reaching the BP goal of < 140/90 mmHg or < 130/80 mmHg for diabetics were considered as responders. All patients (responders and non-responders) then entered into the titration phase of the study (Phase B):

Second double-blind treatment phase/titration phase (Phase B, from Week 8 to Week 16):

Treatment assignment in the second part of the study was based on the following criteria:

* Responders to Phase A treatment continued to receive the same double-blind treatment for an additional 8 weeks.
* Non-responders Phase A treatment had their treatment assigned as follows:

  * Non-responders to OM 40 mg were treated with OM/HCTZ 40/12.5 mg for an additional 8 weeks.
  * Non-responders to OM/HCTZ 40/12.5 mg were uptitrated to OM/HCTZ 40/25 mg for an additional 8 weeks. During Phase B of the study, visits were held 12 and 16 weeks after randomisation (Visits 5 and 6, respectively).

The study ended at Visit 6 and a final examination was performed. A safety follow-up (SFU) telephone contact was performed 2 weeks after the end of the treatment. An SFU visit was performed if deemed necessary by the investigator.

Sphygmomanometer was used for BP measurement throughout the trial. BP was measured at all visits as nearly as possible at the same time of the day as trough readings (24 ± 2 h after last drug intake) after a 10 minute rest period. Three separate sitting BP measurements were taken at least 1 minute apart from each other. The 3 results were then averaged and rounded to a whole integer.

Patients with sBP values > 200 mmHg and/or dBP values > 120 mmHg at any time during the study were to be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of essential hypertension, either treatment-naive or including currently on anti-hypertensive medication (in Italy only treatment naive patients) in whom it is medically justifiable to withdraw treatment , and who are likely to meet the required BP inclusion criteria at randomisation:

  * Mean sitting dBP ≥ 100 mmHg and ≤ 120 mmHg.
  * Mean sitting sBP ≥ 160 mmHg and ≤ 200 mmHg.

Main Exclusion Criteria:

* Mean sitting sBP values > 200 mmHg and/or dBP > 120 mmHg.
* Pregnant or nursing women.
* Patients with serious disorders which may limit the ability to evaluate the efficacy or safety of the tested medication, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine or metabolic, haematological, oncological, neurological, and psychiatric diseases. The same applies for immunocompromised and/or neutropenic patients.
* Patients with secondary hypertension of any aetiology such as renal disease, pheochromocytoma, or Cushing's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Fogari, MD, Principal Investigator — Medical Clinic Policlinico San Matteo University of Pavia Italy
Locations (65):
- Croatia (6):
  - Rijeka
  - Slavonski Brod
  - Split
  - Varaždin
  - Zadar
  - Zagreb
- Czechia (10):
  - Benátky nad Jizerou
  - Bílovec
  - Brodce
  - Jablonec nad Nisou
  - Mladá Boleslav
  - Prague
  - Rokycany
  - Tábor
  - Teplice
  - Uničov
- Denmark (3):
  - Aalborg
  - Ballerup Municipality
  - Vejle
- Germany (16):
  - Berlin
  - Cologne
  - Dresden
  - Einbeck
  - Essen
  - Giengen an der Brenz
  - Großheirath
  - Hamburg
  - Hanau
  - Heidelberg
  - Künzing
  - Leipzig
  - Lollar
  - Mannheim
  - München
  - Nuremberg
- Israel (9):
  - Ashkelon
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Petah Tikva
  - Tel Aviv
  - Tel Litwinsky
- Italy (8):
  - Busto Arsizio
  - Ferrara
  - Pavia
  - Pisa
  - San Daniele del Friuli
  - Sassari
  - Somma Lombardo
  - Venezia
- Poland (7):
  - Bialystok
  - Gdansk
  - Gdynia
  - Lublin
  - Płock
  - Warsaw
  - Wąbrzeżno
- Romania (6):
  - Baia Mare
  - Brăila
  - Bucharest
  - Cluj-Napoca
  - Oradea
  - Suceava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fogari R, Taddei S, Holm-Bentzen M, Baszak J, Melani L, Schumacher K. Efficacy and safety of olmesartan medoxomil 40 mg/hydrochlorothiazide 12.5 mg combination therapy versus olmesartan medoxomil 40 mg monotherapy in patients with moderate to severe hypertension: a randomized, double-blind, parallel-group, multicentre, multinational, phase III study. Clin Drug Investig. 2010;30(9):581-97. doi: 10.2165/11536710-000000000-00000. PMID 20593911

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the arms OM 40 mg and OM/HCTZ 40/12.5 mg, respectively in Phase A are the same ones who started, depending on being a responder or non-responder in the arms of Phase B continuing with OM 40 mg and OM/HCTZ 40/12.5 mg or uptitration to OM/HCTZ 40/12.5 mg and OM/HCTZ 40/25, respectively of Phase B.
Groups:
- Phase A/OM 40: Olmesartanmedoxomil (OM)40 mg tablets. OM 40: Initially patients were to be treated with Olmesartanmedoxomil (OM)40 mg tablets once daily for 8 weeks. After 8 weeks non-responders were to be uptitrated to OM/HCTZ 40/12.5 mg and responders remained on the previous therapy for further 8 weeks.
- Phase A/OM/HCTZ 40/12.5: Olmesartanmedoxomil (OM) /Hydrochlorothiazide (HCTZ)40/12.5 mg tablets. OM/HCTZ 40/12.5: Initially patients were to be treated with Olmesartanmedoxomil (OM) /Hydrochlorothiazide (HCTZ)40/12.5 mg tablets once daily for 8 weeks. After 8 weeks non-responders were to be uptitrated to OM/HCTZ 40/25 mg and responders remained on the previous therapy for further 8 weeks.
- Phase B/ OM 40 mg Responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Responders to OM 40 mg treatment were to continue treatment with OM 40 mg.
- Phase B/ OM 40 mg Non-responder: Phase B (second double-blind treatment phase, 8 weeks duration):
  Non-responders to OM 40 mg treatment were to be up-titrated to OM/HCTZ 40/12.5 mg.
- Phase B OM/HCTZ 40/12.5 mg Responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Responders to OM/HCTZ 40/12.5 mg treatment were to continue treatment with OM/HCTZ 40/12.5 mg.
- Phase B/ OM/HCTZ 40/12.5 mg Non-responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Non-responders to OM/HCTZ 40/12.5 mg treatment were to be up- titrated to OM/HCTZ 40/25 mg.
Period: Phase A: Randomization to Week 8
Arm/Group | Phase A/OM 40 | Phase A/OM/HCTZ 40/12.5 | Phase B/ OM 40 mg Responders | Phase B/ OM 40 mg Non-responder | Phase B OM/HCTZ 40/12.5 mg Responders | Phase B/ OM/HCTZ 40/12.5 mg Non-responders
Started | 285 | 561 | 0 | 0 | 0 | 0
Completed | 268 | 524 | 0 | 0 | 0 | 0
Not Completed | 17 | 37 | 0 | 0 | 0 | 0
Period: Phase B: Week 8 to Week 16
Arm/Group | Phase A/OM 40 | Phase A/OM/HCTZ 40/12.5 | Phase B/ OM 40 mg Responders | Phase B/ OM 40 mg Non-responder | Phase B OM/HCTZ 40/12.5 mg Responders | Phase B/ OM/HCTZ 40/12.5 mg Non-responders
Started | 0 | 0 | 129 | 139 | 336 | 188
Completed | 0 | 0 | 128 | 137 | 333 | 186
Not Completed | 0 | 0 | 1 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OM 40 | OM/HCTZ 40/12.5 | Total
Number analyzed (Participants) | 285 | 561 | 846
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 211 | 454 | 665
  >=65 years | 74 | 107 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (11.46) | 55.5 (10.57) | 55.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 267 | 395
  Male | 157 | 294 | 451
Trough Sitting dBP [Mean (Standard Deviation); unit: mmHg] — Sitting diastolic blood pressure at baseline
  mmHg | 104.5 (4.0) | 104.6 (4.2) | 104.6 (4.1)
Trough Sitting sBP [Mean (Standard Deviation); unit: mmHg] — Sitting systolic blood pressure
  mmHg | 168.0 (7.7) | 168.5 (8.4) | 168.3 (8.1)
Body Mass Index [Mean (Standard Deviation); unit: kg.m^2] | 29.64 (4.8) | 29.17 (4.665) | 29.35 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: dBP Change After 8 Weeks Phase A
Description: Reduction in Mean Trough Sitting dBP (mmHg) from Baseline (Week 0) to Week 8
Time Frame: Eight weeks
Measure: Mean (Standard Deviation); unit: mmHG
Groups:
- OM 40: Olmesartanmedoxomil (OM)40 mg tablets. OM 40: Initially patients were to be treated with Olmesartanmedoxomil (OM)40 mg tablets once daily for 8 weeks.
- OM/HCTZ 40/12.5: Olmesartanmedoxomil (OM) /Hydrochlorothiazide (HCTZ)40/12.5 mg tablets. OM/HCTZ 40/12.5: Initially patients were to be treated with Olmesartanmedoxomil (OM) /Hydrochlorothiazide (HCTZ)40/12.5 mg tablets once daily for 8 weeks.
Arm/Group | OM 40 | OM/HCTZ 40/12.5
Number analyzed (Participants) | 282 | 556
mmHG | -15.8 (9.71) | -18.9 (9.32)
Statistical Analysis 1: Comparison: OM 40 vs OM/HCTZ 40/12.5; Test type: Superiority; p < 0.0001, ANCOVA

2. Primary Outcome: sBP Change After 8 Weeks Phase A
Description: Reduction in Mean Trough Sitting sBP (mmHg) from Baseline (Week 0) to Week 8
Time Frame: Eight weeks
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | OM 40 | OM/HCTZ 40/12.5
Number analyzed (Participants) | 282 | 556
mmHG | -26.5 (14.56) | -31.9 (14.76)
Statistical Analysis 1: Comparison: OM 40 vs OM/HCTZ 40/12.5; Test type: Superiority; p < 0.0001, ANCOVA

3. Secondary Outcome: dBP Change After 8 Weeks Phase B
Description: Reduction in trough sitting diastolic blood pressure after 8 weeks of additional treatment, depending on Phase A treatment and outcome (responder/non-responder).
Time Frame: Eight weeks
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- OM 40 mg Responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Responders to OM 40 mg treatment were to continue treatment with OM 40 mg.
- OM 40 mg Non-responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Non-responders to OM 40 mg treatment were to be up-titrated to OM/HCTZ 40/12.5 mg.
- OM/HCTZ 40/12.5 mg Responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Responders to OM/HCTZ 40/12.5 mg treatment were to continue treatment with OM/HCTZ 40/12.5 mg.
- OM/HCTZ 40/12.5 mg Non-responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Non-responders to OM/HCTZ 40/12.5 mg treatment were to be up- titrated to OM/HCTZ 40/25 mg.
Arm/Group | OM 40 mg Responders | OM 40 mg Non-responders | OM/HCTZ 40/12.5 mg Responders | OM/HCTZ 40/12.5 mg Non-responders
Number analyzed (Participants) | 129 | 139 | 336 | 187
mmHg | -0.5 (6.95) | -9.3 (7.91) | -0.3 (6.68) | -8.0 (8.56)
Statistical Analysis 1: Comparison: OM 40 mg Responders vs OM 40 mg Non-responders vs OM/HCTZ 40/12.5 mg Responders vs OM/HCTZ 40/12.5 mg Non-responders; Test type: Superiority; p < 0.0001, ANCOVA

4. Secondary Outcome: sBP Change After 8 Weeks Phase B
Description: Reduction in trough sitting systolic blood pressure after 8 weeks of additional treatment, depending on Phase A treatment and outcome (responder/non-responder).
Time Frame: Eight weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | OM 40 mg Responders | OM 40 mg Non-responders | OM/HCTZ 40/12.5 mg Responders | OM/HCTZ 40/12.5 mg Non-responders
Number analyzed (Participants) | 129 | 139 | 336 | 187
mmHg | -0.5 (6.95) | -12.4 (11.64) | -0.4 (9.32) | -12.1 (12.69)
Statistical Analysis 1: Comparison: OM 40 mg Responders vs OM 40 mg Non-responders vs OM/HCTZ 40/12.5 mg Responders vs OM/HCTZ 40/12.5 mg Non-responders; Test type: Superiority; p = 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: The study consisted of two sequential phases A and B of 8 weeks duration each.
Description: Adverse events were recorded for all patients who started each of the 2 treatment groups in phase A, as well as in all those patients who, as per their allocation, started the treatment groups in phase B.
Groups:
- Phase B OM/HCTZ 40/12.5 mg Non-responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Non-responders to OM/HCTZ 40/12.5 mg treatment were to be up- titrated to OM/HCTZ 40/25 mg.
- Phase B OM 40 mg Non-responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Non-responders to OM 40 mg treatment were to be up-titrated to OM/HCTZ 40/12.5 mg.
- Phase B OM 40 mg Responders: Phase B (second double-blind treatment phase, 8 weeks duration):
  Responders to OM 40 mg treatment were to continue treatment with OM 40 mg.
- Phase A OM/HCTZ 40/12.5 mg: Phase A (first double-blind treatment phase, 8 weeks duration):
  Arm 2: OM/HCTZ 40/12.5 mg tablet o.d.
- Phase A OM 40 mg: Phase A (first double-blind treatment phase, 8 weeks duration):
  Arm 1: OM 40 mg tablet o.d.
Arm/Group | Phase B OM/HCTZ 40/12.5 mg Non-responders | Phase B OM/HCTZ 40/12.5 mg Responders | Phase B OM 40 mg Non-responders | Phase B OM 40 mg Responders | Phase A OM/HCTZ 40/12.5 mg | Phase A OM 40 mg
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/336 | 0/139 | 0/129 | 0/561 | 0/285
Serious Adverse Events (participants affected / at risk) | 1/188 | 3/336 | 0/139 | 2/129 | 4/561 | 5/285
Other Adverse Events (participants affected / at risk) | 9/188 | 16/336 | 6/139 | 8/129 | 41/561 | 19/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase B OM/HCTZ 40/12.5 mg Non-responders (N=188) | Phase B OM/HCTZ 40/12.5 mg Responders (N=336) | Phase B OM 40 mg Non-responders (N=139) | Phase B OM 40 mg Responders (N=129) | Phase A OM/HCTZ 40/12.5 mg (N=561) | Phase A OM 40 mg (N=285)
Anal fissure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 — Worsening and surgery
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Duodenal ulcer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Brain contusion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Incontinence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Parotid abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Erysipeloid (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 — Erysipel B / Erysipel Crus Left
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase B OM/HCTZ 40/12.5 mg Non-responders (N=188) | Phase B OM/HCTZ 40/12.5 mg Responders (N=336) | Phase B OM 40 mg Non-responders (N=139) | Phase B OM 40 mg Responders (N=129) | Phase A OM/HCTZ 40/12.5 mg (N=561) | Phase A OM 40 mg (N=285)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 9 (9) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 6 (6) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 14 (14) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes